CLINICAL TRIAL: NCT01402674
Title: Long-term Phentermine Pharmacotherapy: An Investigation for Symptoms of Dependence, Cravings, or Withdrawal
Acronym: PC-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Weight Management, California (Other)
Collaborators: American Society of Bariatric Physicians (Other)
Responsible Party: Principal Investigator, Ed J. Hendricks, M.D., Medical Director, Center for Weight Management, California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11061-01
Record Dates: First submitted 2011-07-23; First posted 2011-07-26 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Obesity; Phentermine Withdrawal
Keywords: Obesity treatment; Phentermine; Withholding treatment; Phentermine dependence
MeSH Terms: conditions — Obesity | interventions — Phentermine; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LPT (Active Comparator): Subjects treated with phentermine for 2 years or more.
  Interventions: Drug: Abrupt cessation of phentermine pharmacotherapy
- APT (No Intervention): Patients treated with phentermine for 7 to 14 days.

INTERVENTIONS:
Drug: Abrupt cessation of phentermine pharmacotherapy — Patients will be asked to cease taking phentermine, then to complete psychometric scales 24 and 48 hours later. Patients will be examined at 48 hours by physician who will determine if phentermine should be continued or discontinued.
  Other Names: Phentermine-HCL, generic
  Arms: LPT

SUMMARY:
Phentermine, an amphetamine congener, is the most widely used anti-obesity drug in the U.S. Although phentermine is the agent-of-choice among physicians specializing in obesity treatment, the use of this drug for obesity treatment by other physicians has long been curtailed because misapprehensions regarding phentermine safety. Concerns of phentermine-induced adverse cardiovascular reactions and of phentermine-induced addiction are two fears that have had a profound negative impact on phentermine prescribing. Although warnings of high incidence rates of adverse cardiovascular and psychiatric effects are included in FDA labeling and are often repeated in published reviews, the few clinical reports in the peer-reviewed medical literature of such adverse effects are anecdotal. Fear of phentermine adverse effects does not inhibit the use of phentermine by obesity treatment specialists. A 2008 survey of prescribing practices found that 98% of bariatric medicine specialists used pharmacotherapy in treating obesity and that 97% of those prescribed phentermine as their first choice.

The fear that phentermine has addiction potential appears to be a factor influencing curtailment of use. At the time that phentermine was approved in 1959 the expectations were that it would prove to be addicting, although perhaps less so than amphetamine. These expectations were based on the chemical structural similarities between phentermine and amphetamine and on evidence in rats that phentermine stimulated spontaneous activity. No evidence suggesting the drug had human addiction potential appeared in clinical trials conducted prior to approval.

After 52 years of use there is no evidence in the peer-reviewed medical literature to support the hypothesis that phentermine has significant human addiction potential. Research in addiction medicine has undergone significant development in the last 50 years. Concepts of addiction have shifted from an early focus on tolerance and withdrawal to a current emphasis on the psychological components of dependence. Drug addiction has been redefined as drug dependence and standardized diagnostic criteria have been adopted for drug abuse, dependence and withdrawal. Psychometric testing methods have been developed, validated, and applied clinically for measurements of dependence, drug craving, and withdrawal for a wide variety of substances of abuse including cocaine, heroin, and amphetamine.

Until recently, none of these addiction medicine metrics had been used to study the addiction potential of phentermine. Presumably, since phentermine is an amphetamine congener, any clinical characteristics of dependence or withdrawal should mimic those of amphetamine dependence or withdrawal. One recent retrospective study investigated symptoms occurring when patients treated with long-term phentermine in a weight management program abruptly ceased taking phentermine. The study found that patients on long-term phentermine who ceased phentermine abruptly by their choice did not have an amphetamine-like withdrawal symptom complex. Significantly there was no evidence of phentermine cravings. Further investigation is warranted.

The addiction potential of a drug may be investigated by measuring the drug's propensity to induce dependence, to induce cravings for the drug, and for cessation of the drug to induce characteristic withdrawal symptoms. In the case of amphetamine withdrawal symptoms appear very quickly reaching a maximum at 48 hours after drug cessation.

In this prospective study the addiction potential of phentermine will be assessed with validated psychometric scales to examine patients who have taken phentermine long-term for two years or more. Patients who have taken phentermine for 7 to 14 days will also be assessed. Participating patients who have taken phentermine long-term in this study will be asked to interrupt phentermine therapy for 48 hours to participate in the study. Scale examinations will be conducted at 24 and at 48 hours after drug cessation.

Hypotheses

1. Long-term phentermine-treated (LPT) patients do not develop phentermine dependence or cravings.
2. LPT patients who cease taking phentermine abruptly do not experience amphetamine-like withdrawal symptoms.

Specific Aims

1. To compare the severity of phentermine dependence and craving between LPT patients and acute phentermine-treated (APT) patients
2. To compare the severity of stimulant withdrawal symptoms before and after phentermine cessation in LPT patients.
3. To examine the prevalence of phentermine dependence in LPT patients

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Duration of phentermine treatment

   1. For LPT patients, on phentermine pharmacotherapy consecutively for 2 years or more and willing to take a drug holiday for 48 to 72 hours.
   2. LPT Patients who have taken drug holidays on their own during the most recent 2 years may be included provided there has not been a holiday in the 90 days prior to matriculation in this study.
   3. For APT patients, on phentermine pharmacotherapy for 7 to 14 days at 37.5 mg/day or less.

Exclusion Criteria:

1. Patients with confirmed Axis I psychiatric conditions including depression, ADHD, SAD, bipolar disorder, substance abuse disorders (except caffeine and nicotine) and patients taking drugs for any of these conditions, including anti-depressant drugs, drugs for ADHD and lithium.
2. Patients who were taking phentermine in combination with any other anti-obesity drug.
3. Patients who are taking medications such as beta-blockers, which may modulate the stimulant effect of phentermine.
4. Pregnant patients, nursing mothers, patients with uncontrolled hypertension, hyperthyroidism, severe cardiovascular disease, glaucoma, and known hypersensitivity to phentermine -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Signs or symptoms of phentermine dependence (addiction) | Long-term cohort subjects on phentermine 2 years or more.
  Psychometric scales will be used for assessment of signs or symptoms of phentermine dependence, phentermine withdrawal, or phentermine cravings
Signs or symptoms of phentermine dependence (addiction) | Short-term cohort subjects on phentermine (APT) for 7 to 14 days.
  Psychometric scales will be used for assessment of signs or symptoms of phentermine dependence, or phentermine cravings.

CONTACTS AND LOCATIONS:
Overall Officials: Ed J Hendricks, MD, Principal Investigator — Center for Weight Management
Locations (2):
- United States (2):
  - Center for Weight Management, Roseville, California
  - Center for Weight Management, Sacramento, California

REFERENCES:
- [Background] Hendricks EJ, Greenway FL. A study of abrupt phentermine cessation in patients in a weight management program. Am J Ther. 2011 Jul;18(4):292-9. doi: 10.1097/MJT.0b013e3181d070d7. PMID 20592662
- [Background] Hendricks EJ, Greenway FL, Westman EC, Gupta AK. Blood pressure and heart rate effects, weight loss and maintenance during long-term phentermine pharmacotherapy for obesity. Obesity (Silver Spring). 2011 Dec;19(12):2351-60. doi: 10.1038/oby.2011.94. Epub 2011 Apr 28. PMID 21527891
- [Background] Hendricks EJ, Rothman RB, Greenway FL. How physician obesity specialists use drugs to treat obesity. Obesity (Silver Spring). 2009 Sep;17(9):1730-5. doi: 10.1038/oby.2009.69. Epub 2009 Mar 19. PMID 19300434
- [Background] Kampman KM, Volpicelli JR, McGinnis DE, Alterman AI, Weinrieb RM, D'Angelo L, Epperson LE. Reliability and validity of the Cocaine Selective Severity Assessment. Addict Behav. 1998 Jul-Aug;23(4):449-61. doi: 10.1016/s0306-4603(98)00011-2. PMID 9698974
- [Background] McGregor C, Srisurapanont M, Jittiwutikarn J, Laobhripatr S, Wongtan T, White JM. The nature, time course and severity of methamphetamine withdrawal. Addiction. 2005 Sep;100(9):1320-9. doi: 10.1111/j.1360-0443.2005.01160.x. PMID 16128721
- [Background] McGregor C, Srisurapanont M, Mitchell A, Longo MC, Cahill S, White JM. Psychometric evaluation of the Amphetamine Cessation Symptom Assessment. J Subst Abuse Treat. 2008 Jun;34(4):443-9. doi: 10.1016/j.jsat.2007.05.007. Epub 2007 Jul 13. PMID 17629443
- [Background] Srisurapanont M, Jarusuraisin N, Jittiwutikan J. Amphetamine withdrawal: I. Reliability, validity and factor structure of a measure. Aust N Z J Psychiatry. 1999 Feb;33(1):89-93. doi: 10.1046/j.1440-1614.1999.00517.x. PMID 10197890
- [Background] Tiffany ST, Singleton E, Haertzen CA, Henningfield JE. The development of a cocaine craving questionnaire. Drug Alcohol Depend. 1993 Dec;34(1):19-28. doi: 10.1016/0376-8716(93)90042-o. PMID 8174499